CLINICAL TRIAL: NCT00001438
Title: A Pilot Study of the Combination of Retinoic Acid and Interferon-Alpha2a for the Treatment of Lymphoproliferative Disorders in Children With Immunodeficiency Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950144; 95-C-0144
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: HIV Infections; Immunologic Deficiency Syndromes; Lymphoproliferative Disorders
Keywords: HIV Infection; Immune Response; Pediatric; Pharmacokinetics; Toxicity
MeSH Terms: conditions — HIV Infections; Immunologic Deficiency Syndromes; Lymphoproliferative Disorders | interventions — Tretinoin; Interferon alpha-2

INTERVENTIONS:
Drug: all-trans-retinoic acid with IFN-alpha2a

SUMMARY:
Patients with congenital or acquired immunodeficiencies are at an increased risk to develop polyclonal or oligoclonal lymphoid malignancies. Some develop a lymphoproliferative disorder that can follow a clinically aggressive course and may represent a pre-malignant lesion. Although most of these lymphoproliferative disorders are of B-cell origin, T-cell or non-B-non-T-cell processes have also been observed. The pathogenesis is only partially understood.

In the case of pre-malignant conditions it is often difficult to know when and whether a therapeutic intervention is necessary and a careful consideration of potential treatment-associated morbidity is indicated. Therapies have ranged from influencing the possible infectious etiology (by treating with acyclovir), decreasing the amount of immunosuppression (in transplant patients), to the use of immunomodulatory agents, including interferons and interleukins. Recent data have indicated that the use of differentiating agents, such as the retinoids, might offer yet another treatment option. In the current study we will try to get a better understanding of the pathogenesis and natural course of lymphoproliferative disorders in immunodeficient children.

The study will have two parts: an initial observation period to obtain information on the natural course of these disorders, and then a six month treatment period with the combination of a differentiating agent (13-cis-retinoic acid was used until all-trans-retinoic acid became available on 7/96) with an immunomodulatory agent (interferon-alpha2a, IFN-alpha2a).

DETAILED DESCRIPTION:
Patients with congenital or acquired immunodeficiencies are at an increased risk to develop polyclonal or oligoclonal lymphoid malignancies. Some develop a lymphoproliferative disorder that can follow a clinically aggressive course and may represent a pre-malignant lesion. Although most of these lymphoproliferative disorders are of B-cell origin, T-cell or non-B-non-T-cell processes have also been observed. The pathogenesis is only partially understood. The Epstein-Barr virus (EBV) is thought to play an important role but the human herpes virus type 6 (HHV-6) has been implicated as well. An imbalance in the expression of several cytokines is observed and it is currently not clear whether this sustains the aberrant proliferation or is a result thereof. In the case of pre-malignant conditions it is often difficult to know when and whether a therapeutic intervention is necessary and a careful consideration of potential treatment-associated morbidity is indicated. Therapies have ranged from influencing the possible infectious etiology (by treating with acyclovir), decreasing the amount of immunosuppression (in transplant patients), to the use of immunomodulatory agents, including interferons and interleukins. Recent data have indicated that the use of differentiating agents, such as the retinoids, might offer yet another treatment option. In the current study we will try to get a better understanding of the pathogenesis and natural course of lymphoproliferative disorders in immunodeficient children. The study will mainly be open to children infected with the human immunodeficiency virus but patients who develop a lymphoproliferative disorder post-transplant or as part of another immunodeficiency state may also be enrolled. The study will have two parts: an initial observation period to obtain information on the natural course of these disorders, and then a six month treatment period with the combination of a differentiating agent (13-cis-retinoic acid was used until all-trans-retinoic acid became available on 7/96) with an immunomodulatory agent (interferon-alpha2a, IFN-alpha2a).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Congenital or acquired immunodeficiency (including HIV-1 infection) with a lymphoproliferative disorder (LPD) of any of the following types:

Severe and/or progressive lymphadenopathy with hypergammaglobulinemia.

Diffuse infiltrative lymphocytosis syndrome.

Clinically symptomatic pulmonary lymphoid hyperplasia/lymphocytic interstitial pneumonitis.

Polyclonal B-cell LPD.

No patients with malignant lymphoma.

No active opportunistic infection requiring acute intervention at entry.

THERAPY:

Biologic Therapy:

At least 30 days since immunomodulating agents or biological response modifiers, e.g.: Interleukin-2, Interferons, Growth hormone, Insulin-like growth factor 1.

Requirement waived for intravenous immunoglobulins for hypogammaglobulinemia.

Concurrent post-transplant immunosuppressants allowed. Doses stable for at least 4 weeks prior to entry.

Chemotherapy: At least 30 days since chemotherapy.

Endocrine Therapy:

Concurrent corticosteroids allowed only for lymphocytic interstitial pneumonitis or an autoimmune process. Doses stable for more than 4 weeks prior to entry.

Radiotherapy: At least 30 days since radiotherapy.

Surgery: Not specified.

Antiretroviral therapy (in patients with HIV infection):

Approved anti-HIV medication required.

Initiated at least 8 weeks prior to entry.

Continued throughout protocol treatment.

Prophylaxis for Pneumocystis carinii pneumonia and/or Mycobacterium avium-intracellulare allowed.

Maintenance antifungal or antiviral therapy allowed.

PATIENT CHARACTERISTICS:

Age: Under 18.

Performance status: Not specified.

One or more of the following laboratory findings (within 4 weeks of starting retinoic acid and interferon-alpha , and which have not resolved within 2 weeks of starting):

Creatinine greater than 2 times the upper limit of normal;

Liver transaminases greater than 5 times the upper limit of normal (children with chronically elevated liver enzymes with a proven etiology can be enrolled, but will not be evaluable for liver toxicity); or

Bilirubin greater than 3 times the upper limit of normal.

Patients receiving treatment for an acute infection must have completed therapy at least 14 days prior to starting therapy with retinoic acid and interferon-alpha.

OTHER:

Able to swallow capsules.

No requirement for drugs suspected of causing pseudotumor cerebri for which alternatives cannot be substituted, e.g.: Tetracycline, Nalidixic acid, Nitrofurantoin, Phenytoin, Lithium, Amiodarone, Vitamin A (except as a multivitamin supplement component).

No critical or clinically unstable illness.

No pregnant or nursing women.

Effective contraception encouraged in fertile patients.

Parent or legal guardian available to give informed consent and deemed sufficiently reliable to return for followup visits.

No critically ill or critically unstable children.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1995-06; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sidell N, Taga T, Hirano T, Kishimoto T, Saxon A. Retinoic acid-induced growth inhibition of a human myeloma cell line via down-regulation of IL-6 receptors. J Immunol. 1991 Jun 1;146(11):3809-14. PMID 2033252
- [Background] Su IJ, Cheng AL, Tsai TF, Lay JD. Retinoic acid-induced apoptosis and regression of a refractory Epstein-Barr virus-containing T cell lymphoma expressing multidrug-resistance phenotypes. Br J Haematol. 1993 Dec;85(4):826-8. doi: 10.1111/j.1365-2141.1993.tb03235.x. PMID 7918055
- [Background] Aviles A, Diaz-Maqueo JC, Garcia EL, Talavera A, Guzman R. Maintenance therapy with interferon alfa 2b in patients with diffuse large cell lymphoma. Invest New Drugs. 1992 Nov;10(4):351-5. doi: 10.1007/BF00944195. PMID 1487412